CLINICAL TRIAL: NCT06165848
Title: Effects Of Different Anesthesia Applications On Mood, Depression, And Anxiety Levels In Burn Patients
Status: Completed | Type: Observational
Sponsor: T.C. Sağlık Bakanlığı Ankara Bilkent Şehir Hastanesi (Other)
Responsible Party: Sponsor
Other Study IDs: 11260011; Ayça Tuba Dumanlı Özcan (Other: Ankara Şehir Hastanesi, Anesteziyoloji ve Reanimasyon); Betül Akaycan (Other: Ankara Şehir Hastanesi, Psikiyatri); Serdar Süleyman Can (Other: Ankara Şehir Hastanesi, Psikiyatri); Özlem Karakaya (Other: Ankara Şehir Hastanesi, Psikiyatri); Emine Sönmez (Other: Ankara Şehir Hastanesi, Anesteziyoloji ve Reanimasyon)
Record Dates: First submitted 2023-08-20; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Burn Unspecified Degree; Deep Sedation
Keywords: Burn patient; Depression; Ketamine; Suicidal tendencies
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General anesthesia: After preoxygenation, anesthesia induction was performed with 2 mg/kg IV propofol and 1 mcg/kg IV fentanyl in the general anesthesia group. Anesthesia was maintained with a mixture of 0.3-0.5 mcg/kg/min remifentanil, 2% sevoflurane, 50% air, 50% oxygen. The Montgomery-Asberg Depression Rating Scale (MADRS), the Hamilton Anxiety Rating Scale (HAM-A), and the Beck Scale for Suicide Ideation (BSSI) were administered preoperatively and on postoperative day one by a psychiatrist.
- Sedation anesthesia: In the sedation group, 1 mcg/kg IV fentanyl and 1 mg/kg IV ketamine were administered at induction, and 30-50 mg IV propofol was added if necessary to maintain anesthesia. The Montgomery-Asberg Depression Rating Scale (MADRS), the Hamilton Anxiety Rating Scale (HAM-A), and the Beck Scale for Suicide Ideation (BSSI) were administered preoperatively and on postoperative day one by a psychiatrist.

SUMMARY:
Adequate and effective pain management and prevention of depression are essential in burn patients. This study aims to investigate the effects of ketamine sedation in burn patients in terms of mood disorders, depression, anxiety, and suicidal tendency during intensive care follow-up in the postoperative period.

DETAILED DESCRIPTION:
Aim: Adequate and effective pain management and prevention of depression are essential in burn patients. This study aims to investigate the effects of ketamine sedation in burn patients in terms of mood disorders, depression, anxiety, and suicidal tendency during intensive care follow-up in the postoperative period.

Methods: The study was conducted with 67 patients between 18 and 65 years of age, who were ASA I-II class, had basic communication skills, no previous diagnosis of psychiatric illness, and no history of neuropsychiatric or cognitive disease or related treatment. After preoxygenation, anesthesia induction was performed with 2 mg/kg IV propofol and 1 mcg/kg IV fentanyl in the general anesthesia group. Anesthesia was continued with a mixture of 0.3-0.5 mcg/kg/min remifentanil, 2% sevoflurane, 50% air, 50% oxygen. In the sedation group, 1 mcg/kg IV fentanyl and 1 mg/kg IV ketamine were administered at induction; anesthesia was maintained by adding 30-50 mg IV propofol if necessary. The Montgomery-Asberg Depression Rating Scale (MADRS), the Hamilton Anxiety Rating Scale (HAM-A), and the Beck Scale for Suicide Ideation (BSSI) were administered preoperatively and on postoperative day one by the psychiatrist.

ELIGIBILITY:
Inclusion Criteria:

* Who were ASA I-II class,
* Had basic communication skills,
* No previous diagnosis of psychiatric illness,
* No history of neuropsychiatric or cognitive disease or related treatment.

Exclusion Criteria:

* With a previous diagnosis of psychiatric illness,
* Neuropsychiatric or cognitive illness,
* Or a history of related treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes aged 18 to 65 years will be included in the study.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS), | 72 hours
  In order to determine whether there is negative mood and depression; Montgomery-Asberg Depression Rating Scale (MADRS) was administered by the psychiatrist .
Hamilton Anxiety Rating Scale (HAM-A) | 72 hours
  For anxiety; Hamilton Anxiety Rating Scale (HAM-A) was administered by the psychiatrist .
Beck Suicidal Ideation Scale (BSSI) | 72 hours
  To determine whether there is suicidal ideation; Beck Suicidal Ideation Scale (BSSI) was administered by the psychiatrist .

CONTACTS AND LOCATIONS:
Overall Officials: Ayça Tuba Özcan, Principal Investigator — Ankara Bilkent Şehir Hastanesi
Locations (1):
- Ankara Bilkent Şehir Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: 10 years

REFERENCES:
- [Result] Phillips JL, Norris S, Talbot J, Birmingham M, Hatchard T, Ortiz A, Owoeye O, Batten LA, Blier P. Single, Repeated, and Maintenance Ketamine Infusions for Treatment-Resistant Depression: A Randomized Controlled Trial. Am J Psychiatry. 2019 May 1;176(5):401-409. doi: 10.1176/appi.ajp.2018.18070834. Epub 2019 Mar 29. PMID 30922101
- [Result] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Result] Phillips JL, Norris S, Talbot J, Hatchard T, Ortiz A, Birmingham M, Owoeye O, Batten LA, Blier P. Single and repeated ketamine infusions for reduction of suicidal ideation in treatment-resistant depression. Neuropsychopharmacology. 2020 Mar;45(4):606-612. doi: 10.1038/s41386-019-0570-x. Epub 2019 Nov 23. PMID 31759333